CLINICAL TRIAL: NCT00003789
Title: A Randomized Phase III Trial of Hyperthermic Isolated Limb Perfusion and Melphalan With and Without Tumor Necrosis Factor in Patients With Localized Advanced Extremity Melanoma
Brief Title: Melphalan With or Without Tumor Necrosis Factor in Treating Patients With Locally Advanced Melanoma of the Arm or Leg
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01843; Z0020; ACOSOG-Z0020; CDR0000066929; NCI-03-C-0137; U10CA076001 (NIH); NCT00056732 (obsolete NCT alias)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-07-16 (Estimated); Status verified 2013-06

CONDITIONS: Recurrent Melanoma; Stage III Melanoma
MeSH Terms: conditions — Melanoma | interventions — Melphalan; Tumor Necrosis Factors; Tumor Necrosis Factor-alpha

ARMS (2):
- Arm I (Experimental): Patients undergo hyperthermic isolated perfusions of the lower limb by either the external iliac vessels or the common femoral vessels. Patients undergo perfusions of the upper extremity by the axillary artery and vein using an infraclavicular/axillary incision. Melphalan is introduced into the perfusion by slow injection over 5 minutes and allowed to remain for a total of 60 minutes.
  Interventions: Drug: isolated limb perfusion; Drug: melphalan; Other: pharmacological study; Other: laboratory biomarker analysis
- Arm II (Experimental): Patients undergo hyperthermic isolated perfusions as in arm I. Tumor necrosis factor is administered by slow injection into the arterial line and allowed to remain for a total of 90 minutes. Melphalan is introduced into the perfusion as in arm I and allowed to remain for a total of 60 minutes.
  Interventions: Drug: isolated limb perfusion; Biological: recombinant tumor necrosis factor family protein; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: isolated limb perfusion — Undergo isolated limb perfusion
  Other Names: isolated limb infusion
Drug: melphalan — Given via limb perfusion
  Other Names: Alkeran; CB-3025; L-PAM; L-phenylalanine mustard; L-Sarcolysin
  Arms: Arm I
Biological: recombinant tumor necrosis factor family protein — Given via slow injection into the arterial line
  Other Names: tumor necrosis factor; Tumor Necrosis Factor Family Protein
  Arms: Arm II
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Randomized phase III trial to compare the effectiveness of hyperthermic isolated limb perfusion of melphalan with or without tumor necrosis factor in treating patients who have locally advanced melanoma of the arm or leg. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Heating melphalan to several degrees above body temperature and infusing it only to the area around the tumor may kill more tumor cells. It is not yet known whether combining melphalan with tumor necrosis factor is more effective than melphalan alone in treating melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Compare hyperthermic isolated limb perfusion with melphalan with or without tumor necrosis factor, in terms of response proportion for lesions in the perfusion field, in patients with locally advanced extremity melanoma.

II. Compare the local recurrence-free survival, improvement in regional symptoms related to tumor, and overall survival in patients treated with these regimens.

III. Compare the toxicity of these regimens in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to tumor burden (high vs low), prior reperfusion (melphalan vs other), regional nodal site (yes vs no), and participating center. Patients are randomized to one of two treatment arms.

ARM I: Patients undergo hyperthermic isolated perfusions of the lower limb by either the external iliac vessels or the common femoral vessels. Patients undergo perfusions of the upper extremity by the axillary artery and vein using an infraclavicular/axillary incision. Melphalan is introduced into the perfusion by slow injection over 5 minutes and allowed to remain for a total of 60 minutes.

ARM II: Patients undergo hyperthermic isolated perfusions as in arm I. Tumor necrosis factor is administered by slow injection into the arterial line and allowed to remain for a total of 90 minutes. Melphalan is introduced into the perfusion as in arm I and allowed to remain for a total of 60 minutes.

Patients are followed within 6 weeks, at 3, 6, and 12 months, every 6 months for 4 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven locally advanced melanoma of an extremity

  * One or more evaluable in-transit metastases
  * All disease within the perfusion field of the extremity (with no local resection options short of amputation)
  * Disease outside of perfusion field (with no local resection options short of amputation) if all the following are true:

    * High tumor burden (more than 10 lesions or any single lesion greater than 3 cm)
    * Presence of pain, edema, skin breakdown, or decreased mobility
    * Greater than 80% of known tumor is within extremity perfusion field
    * Life expectancy more than 6 months
    * No brain metastases
* At least 1 bidimensionally measurable lesion
* Patients who received prior prophylactic isolated limb perfusion (ILP) must have 1 of the following:

  * Disease-free interval for at least 6 months after prior ILP with melphalan
  * Disease-free interval for at least 3 months after prior ILP with an agent other than melphalan
* Patients who received prior therapeutic ILP must have 1 of the following:

  * Partial response of at least 3 months duration after prior ILP with melphalan
  * Stable response or disease progression after ILP without melphalan (performed at least 3 months prior to study)
* Performance status - ECOG 0-2
* Performance status - Zubrod 0-2
* See Disease Characteristics
* Platelet count at least 100,000/mm^3
* WBC greater than 2,500/mm^3
* Hemoglobin greater than 9 g/dL
* Bilirubin less than 1.25 times ULN
* AST and ALT less than 2 times ULN
* Alkaline phosphatase less than 2 times ULN
* Coagulation studies normal or within 1 second of upper limit of normal (ULN)
* Creatinine less than 1.5 mg/dL
* Creatinine clearance greater than 50 mL/min
* Calcium less than 12 mg/dL
* No severe peripheral vascular disease (claudication or other ischemic peripheral vascular disease [e.g., venous thrombosis or occlusive peripheral arterial disease])
* No New York Heart Association class II-IV heart disease (congestive heart failure)
* No uncontrolled or life-threatening cardiac arrhythmia
* No myocardial infarction within the past year
* No unstable angina
* No symptomatic cerebral or carotid artery disease
* No pulmonary embolism within the past year
* Other prior malignancy allowed if completed curative therapy, disease-free for at least 5 years, and at low risk for recurrence
* No active peptic ulcer disease within the past year
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No known melphalan hypersensitivity
* No known hypersensitivity to any component of tumor necrosis factor alpha formulation
* No contraindications to ionotropic agents (e.g., dopamine or neosynephrine)
* No concurrent infections uncontrolled with antibiotics
* HIV negative
* At least 1 month since prior biologic therapy
* See Disease Characteristics
* At least 1 month since prior chemotherapy
* At least 4 months since prior isolated limb perfusion
* At least 1 month since prior radiotherapy
* See Disease Characteristics
* At least 12 months since prior coronary artery surgery or angioplasty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 1999-03; Primary Completion 2004-01 (Actual)

PRIMARY OUTCOMES:
CR proportion | Up to 3 months after completion of study treatment
  Response will be calculated based on the 3-month follow-up assessment of presence of absence of complete response. This will be done using the logistic regression model.
Incidence of adverse events, graded according to NCI CTC version 2.0 | Up to 1 month after completion of study treatment
  The quantification and between-arm comparison of toxicity will be studied.

SECONDARY OUTCOMES:
Local progression-free survival | Up to 12 years
  Time to event outcome models will be based on proportional hazard regression.
Overall survival | Up to 12 years
  Time to event models will be based on proportional hazard regression.

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Fraker, Principal Investigator — American College of Surgeons
Locations (1):
- American College of Surgeons Oncology Group, Durham, North Carolina, United States